CLINICAL TRIAL: NCT06375096
Title: Bone Mineral Density in Children With Graves' Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadeer Youssef Mahmoud Nasr, Bone mineral density in children diagnosed with graves' disease, Assiut University
Other Study IDs: Graves' disease
Record Dates: First submitted 2024-03-25; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Bone Density, Low; Bone Mineral Density in Children With Graves' Disease
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: evaluate bone mineral density — observation effect of graves' in bone mineral density in children

SUMMARY:
to evaluate bone mineral density in children with graves' disease

ELIGIBILITY:
Inclusion Criteria:

* age at enrollment ≥2 years to < 18 years
* both sexes
* the patients should be diagnosed with graves'

Exclusion Criteria:

* patients less than 2 years
* patients more than 18 years
* Controlled GD patients on antithyroid
* patients with other endocrine diseases

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children diagnosed with graves' disease, more than 2 years and less than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
bone mineral density | 1 month
  measure bone mineral density in children diagnosed with graves' disease, to evaluate the effect of the disease on it and the effect of antithyroid medication after that

IPD SHARING:
Plan to Share IPD: Undecided